CLINICAL TRIAL: NCT03105726
Title: Medical Care Versus Ventricular Assist Device in Patients With NYHA Class IV Congestive Heart Failure: a Non Randomized Comparison of Clinical and Economic Outcomes
Brief Title: Medical Care Versus Ventricular Assist Device for the Management of End-stage Heart Failure (MEVADE)
Acronym: MEVADE
Status: Completed | Type: Observational
Sponsor: Joe Elie Salem (Other)
Responsible Party: Sponsor-Investigator, Joe Elie Salem, MD, PhD, Groupe Hospitalier Pitie-Salpetriere
Organization: Groupe Hospitalier Pitie-Salpetriere (Other)
Other Study IDs: C-1421-14-05
Record Dates: First submitted 2017-04-04; First posted 2017-04-10 (Actual); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Heart Failure; Heart Transplantation; Heart-Assist Devices
Keywords: End Stage Heart Failure; New York Heart Association functional class III or IV; Heart transplantation; Ventricular assisted devices; Cardiogenic shock
MeSH Terms: conditions — Heart Failure; Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group I: Group managed by ventricular assist devices in first intention in Bad-Oeynhausen, Germany
- Group II: Group managed with medical therapy, heart transplantation, or both, in first intention,in Paris, France

SUMMARY:
End-stage heart failure (ESHF) represents a major burden in terms of quality of life, mortality and costs. The current practice in France is to treat patients with ESHF by a combination of drugs and lifestyle interventions before proposing heart transplant (HT) if there is no contraindication. In the Heart and Diabetes Center of Bad Oyenhausen (BO) in Germany, patients presenting with ESHF are preferentially managed by ventricular assist device (VAD) therapy. The primary purpose of this study was to compare the outcomes of these two strategies in the management of ESHF and associated consumption of resources.

ELIGIBILITY:
Inclusion Criteria: All patients presenting with end-stage heart failure defined as:

* A left ventricular ejection fraction ≤25%
* Or an oxygen consumption peak < 14 mL/kg/min
* Or severe symptoms (NYHA class III or IV) despite optimal medical treatment
* Or a cardiogenic shock

Exclusion Criteria:

* Age over 70 years
* Active neoplasia
* Suspected or active systemic infection
* Body mass index ≥40 kg/m2
* Severe chronic obstruction pulmonary disease
* Evidence of intrinsic hepatic diseases defined as liver enzyme values ≥ 5 times the upper limit of normal within 4 days before the randomisation, or biopsy proven liver cirrhosis
* Significant chronic renal impairment with persistent creatinine >2.5 or clearance < 25ml/min
* Pregnant or lactating female
* Patient under consideration for conventional revascularization procedures, therapeutic valvular repair, left ventricular procedure or cardiomyoplasty
* Presence of implanted mechanical aortic valve that will not be converted to bioprothesis at the time of ventricular assist device implantation
* Evidence of intrinsic hepatic diseases defined as liver enzyme values ≥ 5 times the upper limit of normal, or biopsy proven liver cirrhosis
* Occurrence of stroke within 90 days or history of cerebrovascular disease with major (≥ 80%) extracranial or carotid stenosis documented by Doppler study
* Confirmation by neurologist of impairment of cognitive function, presence of Alzheimer's disease or any other form of irreversible dementia or both
* Major peripheral vascular disease accompanied by pain on rest or leg ulceration
* Recent history of psychiatric disease that is likely to impair compliance
* Drug or alcohol dependence
* Difficult social surroundings

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients presenting with end-stage heart failure between November 2010 and October 2011 at the Heart and Diabetes Center of Bad Oeynhausen, and who underwent ventricular assist device implantations were included in group I. All patients presenting with end-stage heart failure to the Hôpital Européen Georges Pompidou or the Groupe Hospitalier Pitié-Salpêtrière, during that same period, were included in group II.
Sampling Method: Non-Probability Sample
Enrollment: 224 (Actual)
Dates: Start 2010-11 (Actual); Primary Completion 2013-10 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Survival | two years
  The primary outcome was comparison of survival at two years between the two treatment strategies

SECONDARY OUTCOMES:
Resource consumption | Two years
  One secondary outcomes was comparison of the treatment strategies up to two years of follow-up about resource consumption.
Costs | Two years
  One secondary outcomes was comparison of the treatment strategies up to two years of follow-up about costs.
Costs versus survival | Two years
  One secondary outcomes was comparison of the treatment strategies up to two years of follow-up about costs versus survival.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle IDZ Durand-Zaleski, MD, PhD, Study Director — UMRS 1123, Unité de Recherche Clinique en Économie de la Santé, Ile de France Hôpital Hôtel Dieu, Santé Publique Hôpital Henri Mondor, Paris, France;; Nadia NA Aissaoui, MD, PhD, Principal Investigator — HEGP and Université Paris Descartes; Jan JG Gummert, M.D, PhD, Study Chair — Herz und Diabetes Zentrum, NRW; Jean-Yves JYF Fagon, MD, PhD, Study Chair

IPD SHARING:
Plan to Share IPD: No